CLINICAL TRIAL: NCT05702775
Title: Endosonography-guided Gallbladder Drainage vs Non-endoscopic Treatment in Patients With Inoperable Acute Cholecystitis: a Multicenter Randomized Clinical Trial (EUS-DRAIN)
Brief Title: Endosonography-guided Gallbladder Drainage vs Non-endoscopic Treatment in Inoperable Acute Cholecystitis
Acronym: EUS-DRAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Miguel Servet (Other)
Responsible Party: Principal Investigator, Jesus Maria Urman Fernandez, Head of Pancreas Unit, Fundacion Miguel Servet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Jesús María Urmán Fernández
Record Dates: First submitted 2022-08-24; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Cholecystitis, Acute
Keywords: Cholecystitis; Non-operable; Endoscopic
MeSH Terms: conditions — Cholecystitis, Acute; Cholecystitis

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, low-intervention, superiority clinical trial with parallel groups for the two treatment strategies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-endoscopic treatment group (Group NE) (No Intervention): Antibiotic treatment will start from the moment of diagnosis in both arms of the study. Following the recommendations of the Clinical Practice Guideline for the Management of Acute Cholecystitis of Tokyo 2018, CAL will be classified into three groups according to severity (I,II,III) and empirical antibiotic treatment will be started according to the recommendations of said guideline
- Endoscopic treatment group (EUS-GBD Group) (Experimental): The procedure will be performed after at least 6 hours of fasting The placement of the drain will be performed using a linear echoendoscope that allows the gallbladder to be punctured from the gastric antrum or the duodenal bulb to generate a cholecystogastrostomy or a cholecystoduodenostomy, respectively. Transmural gallbladder drainage will be performed by placing a metal apposition stent (LAMS) with the 15x15mm Hot AXIOS device (Boston Scientific) in the case of cholecystogastrostomy or 15x10 or 10x10mm in the case of cholecystoduodenostomy.
  Interventions: Procedure: Endoscopic treatment group (EUS-GBD group

INTERVENTIONS:
Procedure: Endoscopic treatment group (EUS-GBD group — The placement of a endoscopic drain performed using a linear echoendoscope that allows the gallbladder to be punctured from the gastric antrum or the duodenal bulb to generate a cholecystogastrostomy or a cholecystoduodenostomy, respectively. Transmural gallbladder drainage will be performed by placing a metal apposition stent (LAMS) with the 15x15mm Hot AXIOS device (Boston Scientific) in the case of cholecystogastrostomy or 15x10 or 10x10mm in the case of cholecystoduodenostomy. Subsequently, the interior of the gallbladder will be irrigated with saline solution until the vesicular content comes out.
  Arms: Endoscopic treatment group (EUS-GBD Group)

SUMMARY:
In this project the investigators propose to carry out a clinical trial that compares non-endoscopic treatment of cholecystitis with antibiotics versus endoscopic drainage in non-operable acute cholecystitism (AC), especially focused on the rate of subsequent EBP and recurrence of AC, as well as the impact on the quality of life, also exploring the costs.

The ultimate goal of this project is to generate knowledge and scientific evidence that makes it easier for health professionals to choose the most appropriate strategy for non-operable patients with lithiasic AC.

Ourworking hypothesis is that endoscopic treatment (EUS-GBD) will significantly reduce the number of EBP compared to non-endoscopic treatment in patients with non-operable lithiasic AC.

DETAILED DESCRIPTION:
Design

* Randomized, open-label, low-intervention, superiority clinical trial with parallel groups for the two treatment strategies.
* Cost study Patients who meet the inclusion criteria and do not meet any exclusion criteria will be invited to participate in the study. Between the formalization of the request and the endoscopic examination, the informed consent will be completed in accordance with Law 41/2002 on patient autonomy without altering the relationship with your doctor or causing any damage to your health.

Patients will be randomized in non-endoscopic group or in endoscopic drainage group.

Antibiotic treatment will start from the moment of diagnosis in both arms of the study. Following the recommendations of the Clinical Practice Guideline for the Management of Acute Cholecystitis of Tokyo 2018.

The duration of antibiotic treatment in undrained patients will be 10 to 14 days as long as the cholecystitis has been cured and it will be 4-7 days after gallbladder drainage (EUS-GBD or PC) as long as the cure has been achieved of cholecystitis.

Endoscopic ultrasound-guided transmural gallbladder drainage (EUS-GBD)will be performed only in the endoscopic treatment arm. The procedure will be performed after at least 6 hours of fasting

* in the first 72 hours after admission
* in a specific endoscopy room with fluoroscopy assistance,
* by endoscopists experienced in endoscopically guided transmural drainage (with experience of more than 25 drainages)
* under direct sedation with propofol The placement of the drain will be performed using a linear echoendoscope that allows the gallbladder to be punctured from the gastric antrum or the duodenal bulb to generate a cholecystogastrostomy or a cholecystoduodenostomy, respectively. Transmural gallbladder drainage will be performed by placing a metal apposition stent (LAMS).

Until the acute cholecystitis is cured, a daily evaluation of the visual analogue pain scale (VAS), temperature measurement and periodic blood tests will be carried out.

All patients will receive regular analgesia. Acute cholecystitis will be considered cured if the patient remains afebrile (<37.5ºC), with controlled abdominal pain and presents normalization or a decrease in the number of leukocytes > 20%.

Antibiotic treatment will be adjusted based on the results of blood cultures (BC) or bile culture if available.

Percutaneous cholecystostomy (PC) need. Those patients included who present sepsis, or a critical clinical situation that do not respond to conservative treatment or that after 72 hours of antibiotic treatment do not present clinical improvement, gallbladder drainage will be considered.

Patients included in the NE group who present these circumstances will undergo a PC. For patients in the EUS-GB group, an attempt will be made to perform EUS-GB drainage as soon as possible, and if this is not possible, drainage will be performed by PC (whose performance does not preclude subsequent EUS-GBD).

Periodic follow-up visits will be carried out: every month and every six months until the end of the follow-up. The visits will preferably be face-to-face, and when this is not possible, they will be carried out by telephone, especially in institutionalized patients or with serious mobility problems.

During these visits,

* Record of complications associated with the treatment received and record of EBP developed since the last visit (especially the presence of biliary colic that did not require admission or assessment in the emergency room). An interview will be conducted to collect the presence of EBP that have not required admission (such as biliary colic or related pain), recording the type and date of appearance.
* In cases of EUS-GBD in which it is decided not to remove the prosthesis, the normal position of the prosthesis will be confirmed by abdominal ultrasound.
* IGICV Gastrointestinal Quality of Life Index Questionnaire
* Monitoring of adverse effects The data collection will be carried out by the principal investigator or the collaborating investigators using a data collection notebook (CRD) anonymously and dissociated from the clinical information by means of a patient identification code. The information will be transferred from the data collection notebook to a database (Redcap). The database will be protected with a password to which only researchers will have access.

The follow-up variables after discharge will be collected during the scheduled visits or through a telephone interview at the first, sixth and twelfth month of follow-up.

The economic variables and costs will be those offered by the economic management units of each center.

Descriptive analysis. For quantitative variables, the arithmetic mean and standard deviation will be calculated (variables that do not follow a normal distribution will be described as median, minimum, maximum, and interquartile range), and categorical variables will be expressed as percentages and their 95% confidence intervals.

An intention-to-treat analysis will be performed regardless of treatment received after randomization.

A per-protocol analysis will also be performed, including only those subjects in each group in whom the assigned treatment is successfully carried out.

Logistic regression techniques will be performed to evaluate possible confounding factors (admission diagnosis, referral center, admission severity, age, sex, follow-up center).

Given that there may be differences in the time to recurrence in both groups, we will also assess the appearance of recurrences using Cox risk regression models.

Patients will be censored at the time of loss to follow-up or death. Any urgent admission for biliary complications will be considered as an EBP.

The study data will initially be dissociated from the identity of the participant, by means of an ID, by the responsible physician. The relationship between the ID and the identity of the participant will be kept by the research doctors in a file protected with a personal password.

The data will be entered into the database anonymously with the participant's ID, to maintain their anonymity. The database will be password protected and only accessible by researchers.

Patients eligible for our study will undergo an informative interview with a member of the research team, in which the objectives of the study will be explained, permission will be requested for their inclusion in the study, and informed consent will be given for their inclusion. With the acceptance by the patient and the signing of the informed consent.

The benefit for patients that we are looking for with this study is to significantly reduce the risk of readmission due to EBP in patients with acute lithiasic cholecystitis who are not candidates for surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years.
* Definitive diagnosis of acute lithiasic cholecystitis according to the GP Tokyo 2018 criteria.
* Surgical decision of inoperable patient (if one or more of the following criteria is met: age ≥80 years, American Society of Anesthesiology (ASA) III or more, Charlson Comorbidity Index > 5 and/or Karnofsky < 50 or decision of the patient not to have surgery.
* Signature of the informed consent of the study

Exclusion Criteria:

* Operable acute cholecystitis.
* Refusal of the patient to participate in the study.
* Anatomy of the GI tract altered by previous hepatobiliary or upper GI surgery.
* Ascites.
* Inability to tolerate endoscopy sedation, perforation of the digestive tract, or other contraindication to endoscopy.
* Patients with decompensated cirrhosis, portal hypertension and/or gastric varices
* Coagulopathy with uncorrectable INR>1.5 or thrombocytopenia <50,000/mm3 uncorrectable.
* Other diagnoses on admission (choledocholithiasis, liver abscesses, acute pancreatitis or biliopancreatic neoplasia).
* Hemodynamic instability.
* Baseline ECOG >=4
* Survival expectancy < 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative rate of biliopancreatic events development at one year of follow-up | 2 years
  Biliopancreatic event (BPE): event related to biliary pathology such as acute cholecystitis, acute cholangitis, symptomatic choledocholithiasis, acute pancreatitis mild-moderate, severe acute pancreatitis, biliary colic (complicated or uncomplicated), liver abscess

SECONDARY OUTCOMES:
Proportion of technical success of EUS-GBD and the complications | 2 years
  Describe the proportion of technical success of EUS-GBD and the complications associated with the management of the patients included in the study
Evaluate healing and time to healing of acute cholecystitis | 2 years
  Evaluate healing and time to healing of acute cholecystitis
Evaluate the duration of the index admission | 2 years
  Evaluate the duration of the index admission
Evaluate the duration of antibiotic treatment | 2 years
  Evaluate the duration of antibiotic treatment
Evaluate the need for percutaneous cholecystostomy | 2 years
  Describe the need for percutaneous cholecystostomy in both groups
Evaluate mortality during admission and follow-up in the two treatment groups | 2 years
  Evaluate mortality during admission and follow-up in the two treatment groups
Evaluate the costs of the two treatment strategies: hospital costs of the index admission and the costs generated during the follow-up period related to the biliopancreatic pathology | 2 years
  Evaluate the costs of the two treatment strategies: hospital costs of the index admission and the costs generated during the follow-up period related to the biliopancreatic pathology
Evaluate the digestive symptoms and quality of life of the patients during follow-up | 2 years
  Evaluate the digestive symptoms and quality of life of the patients during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No